CLINICAL TRIAL: NCT06024434
Title: Effects of Specialized Strength Training Protocol On Functional Movement Status of Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RiphahIU Lubna Ali
Record Dates: First submitted 2023-08-26; First posted 2023-09-06 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Sedentary Behavior
Keywords: office workers; functionla movement screening
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise; Walking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental interventional group A (Experimental): Exercises for core, gluts, upper body and lower body
  Interventions: Other: Exercises
- Control group B (Active Comparator): Walking for 30 min 5 days a week
  Interventions: Other: Walking

INTERVENTIONS:
Other: Exercises — Experimental Group Exercises for Core: Crunches, Glute bridges Crunches Glute bridge Week 1-2 (set/rep/sec) Week 3-4 (set/rep/sec) Week 5-6 (set/rep/sec) Exercises for upper body: Push up (4), Bicep curls Exercises Weeks Reps/sets Push up walk out Bicep curls 1-3 16-20*3 Push up Bicep curl with Dumbbell 4-6 12-15*3 Exercises for Lower body: Lunges and Squats Exercises Weeks Reps/set Split Squat with body weight Body weight Squat 1-3 16-20*3 Split Squat with Dumbbell Squat with Dumbbell 4-6 12-15*
  Arms: Experimental interventional group A
Other: Walking — Walking for 30min, 5 days a week
  Arms: Control group B

SUMMARY:
The aim of the study was to determine the effects of specialized strength training protocol on the functional movement status of office workers, and to assess and evaluate the quality of movement patterns and identify any limitations that may exist in order to prevent musculoskeletal injuries, using Functional movement screening. Randomized controlled trials done at Codistan Ventures and Zakori Industries Private Limited. The sample size was 100. The subjects were divided in two groups, 50 subjects in Specialized Strength Training Protocol group and 50 in 30 minute walk group. Study duration was of 6 months. Sampling technique applied was non probability connivance sampling technique. Only 20-35 years office desk workers with no known musculoskeletal deformity were included. Tool used in the study was Functional Movement Screening Test.

DETAILED DESCRIPTION:
As the world is becoming more corporate, the increase in number of hours a person spends in his or her workplace has certainly shifted people towards a sedentary way of life. Sitting and working for a long time in an improper position leads to the tightness and weakness of the muscles, which can lead to musculoskeletal disorders such as neck, shoulders, and lower back pains as well as anatomical disorders such as lordosis, kyphosis, and scoliosis.Most causes of these symptoms include long sitting and excessive leaning. Individuals with areas of muscular weaknesses cannot perform fundamental movement patterns due to compensatory adaptations which can increase the risk of injury. To combat workplace-caused mental and physical exhaustion physical activity has been proven to be an efficient tactic. Physical activity is known not to only treat but prevent the occurrence of a fore coming disease. Being physically active will lead to reduced stress levels and increased productivity. According to World Health Organization facts physical activity refers to all movement including during leisure time, for transport to get to and from places, or as part of a person's work. Both moderate- and vigorous-intensity physical activity improve health that also includes walking for 150-300 minutes a week for adults. Some physical activity is better than doing none. By becoming more active throughout the day in relatively simple ways, people can easily achieve the recommended activity levels.Physical Fitness is defined as the ability to perform physical activity and comprises of components such as flexibility, strength and endurance. A complete physical fitness regimen must target core and extremities. A strong musculoskeletal system is recognized as important component of health related physical fitness. Strength training program provides an opportunity to improve health, physical fitness and quality of life. Core strengthening involving multiplane movements has plausible benefits to improve functional movement patterns. Combination of core strengthening along with upper and lower extremities strengthening program is needed to improve the physical fitness in active individuals to improve their functional status. The topic of FMS (Functional Movement Status) development has received considerable interest owing to the close association between health and well-being, physical activity, and to a lesser degree physical performance.

ELIGIBILITY:
Inclusion Criteria:

Both gender

* Office Workers whose age lies between 15 and 30
* Both male and female gender
* At least 6-8 hours shift per day
* Job duration >6 months
* FMS ≤14

Exclusion Criteria:

reviously diagnosed Musculoskeletal disorder or injury

* Cardiovascular disorders
* Rheumatoid arthritis
* Acute infection

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Functional Movement screening Questionnaire (FMS) | Baseline to 6th week
  FMS is a composite performance measure that is also an injury predictor. it consists of seven basic functional patterns: deep squat, hurdle step, in-line lunge, shoulder mobility, active straight leg raises, trunk stability push-up and rotary stability. each test will be give a score of 3 if performane correct, 2 if performed with compensation, 1 if unable to perform the pattern, 0 if there is pain associated with it. max. score will be 21 and if score is less than 14 that means that person is prone to injury in future.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Care Cloud and Zakori Industries Limited, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No